CLINICAL TRIAL: NCT01675258
Title: Identifying Saliva Markers of Patients With Stomach, Colorectal (Including Pre-cancer Polyp) and Pancreatic Cancers
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Other Study IDs: LSA003-HMO-CTIL
Record Dates: First submitted 2012-08-27; First posted 2012-08-29 (Estimated); Last update posted 2012-08-29 (Estimated); Status verified 2012-07

CONDITIONS: Gastric Cancer; Colorectal Cancer and Pre-cancer Polyps; Pancreatic Cancer
MeSH Terms: conditions — Stomach Neoplasms; Colorectal Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — whole saliva

GROUPS / COHORTS (2):
- Control: Healthy adults above the age of 18 years
  Interventions: Other: Salivary samples
- Study: Adult patients above the age of 18 years with gastric, colorectal (including pre-cancer polyps) or pancreatic cancer
  Interventions: Other: Salivary samples

INTERVENTIONS:
Other: Salivary samples — Each participant will give a sample of saliva through spitting for 10 minutes in a sterile tube.
  Other Names: Salivary Analysis

SUMMARY:
Colorectal cancers account for 783,000 new cases and cause 437,000 deaths per year across the world. Diagnosis in the early stages improves survival rates. Up to now, these cancers are mostly diagnosed only at later stages of the disease's course through histoimmune staining and molecular biology processes on the tissues biopsied from the gastrointestinal system under invasive diagnostic procedures of colonoscopy.

Oral fluid presents a large protein complexity and has been recently used as a diagnostic biofluid for oral, as well as systematic diseases. Using oral fluid as a bio-marker for the colorectal cancer can be advantageous as it contains gastrointestinal fluids, in addition to bacteria and bacteria lysate, which can also serve as a bio-markers' source for colorectal cancers. Proteomic technologies provide the tools needed to discover and identify disease-associated biomarkers.

The aim of the present study is to identify salivary bio-markers in patients suffering from colorectal cancers.

ELIGIBILITY:
Inclusion Criteria:

* Has not yet started treatment for the identified cancer

Exclusion Criteria:

* medically compromised patients
* congenital syndromes
* being treated with radiotherapy or chemotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients identified with gastric, colorectal (including pre-cancer polyps) or pancreatic cancer
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2012-09; Primary Completion 2013-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Moti Moskovitz, DMD, PhD, Principal Investigator — Hadassah Medical Organization; Eyal Shtayer, MD, Principal Investigator — Hadassah Medical Organization; Avi Levin, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Result] Zhang L, Farrell JJ, Zhou H, Elashoff D, Akin D, Park NH, Chia D, Wong DT. Salivary transcriptomic biomarkers for detection of resectable pancreatic cancer. Gastroenterology. 2010 Mar;138(3):949-57.e1-7. doi: 10.1053/j.gastro.2009.11.010. Epub 2009 Nov 18. PMID 19931263